CLINICAL TRIAL: NCT05951348
Title: Comparing Delayed Cord Clamping and Umbilical Cord Milking During Elective Cesarean Section for the Neonatal Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0106748
Record Dates: First submitted 2023-07-06; First posted 2023-07-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-05

CONDITIONS: Umbilical Cord Milking
Keywords: cesarean section; umbilical cord milking; hemoglobin
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate cord clamping (No Intervention): this arm where the patient didn't receive any special maneuver and immediate cord clamping after delivery of the fetus is done
- Delayed cord clamping (Experimental): this arm where the patient receive a delay in cord clamping for 30 seconds after delivery of the fetus
  Interventions: Procedure: Delayed cord clamping for 30 seconds
- Umbilical cord milking (Experimental): this arm where the patient receive stripping of the umbilical cord in the direction of the fetus 10 times in a time frame 10-15 seconds after delivery of the fetus
  Interventions: Procedure: Delayed cord clamping for 30 seconds

INTERVENTIONS:
Procedure: Delayed cord clamping for 30 seconds — waiting for 30 seconds after delivery of the fetus or milking of the cord in the direction of the fetus 10 times in time frame 10-15 seconds
  Other Names: Umbilical cord milking
  Arms: Delayed cord clamping; Umbilical cord milking

SUMMARY:
the study is conducted on the different actions on umbilical cord clamping including immediate cord clamping (ICC) , delayed cord clamping (DCC) for 30 seconds and umbilical cord milking (UCM) for 10-15 seconds in females that are delivered by elective cesarean section , to assess the neonatal outcomes including Hemoglobin and Hematocrit levels after birth in the newborn and the bilirubin level after 72 hrs

DETAILED DESCRIPTION:
the benefit of umbilical cord milking for 10-15 seconds maneuver in cesarean section, that short time can improve the hemoglobin level and prevent anemia in the newborn with improvement of the iron stores for months in infancy without affection on the bilirubin level and the need for phototherapy. This is significant because of the rising rate of cesarean section all over the world make more children are liable for anemia, and by this simple technique it can be prevented.

ELIGIBILITY:
Inclusion Criteria:

* mother's age (20-40) years.
* pregnancy with a healthy singleton
* gestational age of 38-41 0/7 weeks
* uncomplicated pregnancy

Exclusion Criteria

* Any medical or obstetrical complications like hypertension, pre-eclampsia, diabetes any special habits like smoking, and substance abuse
* Rh-negative mothers. The fetal exclusion criteria
* fetus with evidence of intrauterine growth restriction
* infant with serious congenital anomalies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
hemoglobin level | immediately after the intervention
  a blood sample is taken from the umbilical cord of the neonate

SECONDARY OUTCOMES:
bilirubin level | 72 hours after delivery
  trans-cutaneous measurement of the bilirubin level

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer Ahmed Hosny, Alexandria, Egypt